CLINICAL TRIAL: NCT06194773
Title: Evaluation of the Effect of Totalfil and Neosealer Sealers on the Post-endodontic Pain in Mandibular Molars Diagnosed With Symptomatic Irreversible Pulpitis; a Randomized Control Study.
Brief Title: The Effect of Totalfil and Neosealer Sealers on the Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Rania Zaarour, Senior Researcher at Thumbay Research Institute Coordinator, Gulf Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-COD-STD-123-JUNE-2023
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Totalfil (Experimental)
  Interventions: Procedure: Totalfil
- NeoSealer (Experimental)
  Interventions: Procedure: NeoSealer
- AH-Plus (Active Comparator)
  Interventions: Procedure: AH-Plus sealer

INTERVENTIONS:
Procedure: Totalfil — Root canal treatment using TotalFil sealer
  Arms: Totalfil
Procedure: NeoSealer — Root canal treatment using NeoSealer
  Arms: NeoSealer
Procedure: AH-Plus sealer — Root canal treatment using AH-Plus sealer
  Arms: AH-Plus

SUMMARY:
The goal of this clinical trial is to evaluate the effect of Totalfil and Neosealer sealers on post-endodontic pain compared to AH plus sealer in mandibular molars with symptomatic irreversible pulpitis. The main question: do Totalfil and Neosealer sealers affect postoperative pain intensity after root canal treatment in mandibular molars with symptomatic irreversible pulpitis? Participants will undergo root canal treatment using totalfil, Neosealer, or AH-Plus sealer. Researchers will compare Totalfil, Neosealer, and AH-Plus to assess the intensity of post-endodontic pain.

DETAILED DESCRIPTION:
The study will be conducted on 39 mandibular molars; with 13 mandibular mandibular molars in each group (n=13). The patient will be asked to pick an opaque sealed envelope that will contain a number from 1 to 3. The resultant number will determine in which group the participants will be placed. Double blinding will be maintained in this study as the assessor and the patients will not be aware of their group/used root canal sealer.

Group I: Endodontic treatment with obturation using single cone technique with Totalfil sealer.

Group 2: Endodontic treatment with obturation using single cone technique with Neosealer.

Group 3: Endodontic treatment with obturation using single cone technique with AH plus sealer.

Clinical procedure:

1. Patient history will be recorded before starting the procedure.
2. The consent form will be given and signed by the patient.
3. Pre-operative pain will be assessed using VAS.
4. Tooth diagnosis will take place through visualization, percussion, palpation, mobility, electric pulp test as well as cold test before the treatment begins.
5. Pre-operative radiograph will be taken to confirm diagnosis.
6. All the patients will receive local anesthesia: 2% lidocaine with 1:100,000 epinephrine. The inferior alveolar nerve block will be administered.
7. A single tooth will be isolated using a rubber dam, and the access cavity will be prepared using a round bur (no.4) and tapered fissure diamond stone (NO173).
8. The saliva ejector will be introduced below the integrated frame and will be positioned in the corner of the mouth.
9. De-roofing of the pulp chamber will be done using Endo Z bur.
10. After removal of the pulp tissue using an H-file, the working length will be determined with stainless steel hand K-files size #10 and the use of an apex locator and confirmed using intraoral periapical radiographs.
11. All the canals will be prepared using Protaper Gold rotary system using NSK endodontic motor, according to the manufacturer guidelines.
12. To establish apical patency between the files during shaping we will use initial file size #10 between each instrument.
13. Each canal will be irrigated with 30 mL 3% NaOCl and flushed with saline 10 mL between each file during the whole preparation procedure using a plastic syringe with a side vented needle.
14. After completion of cleaning and shaping in all the canals will be flushed with a final rinse of NaOCl, saline and EDTA 17%.
15. For group 1, the canals will be moist and obturated using the single cone technique by gutta percha using Totalfill as a sealer.
16. For group 2, the canals will be moist and obturated using the single cone technique by gutta percha using Neosealer.
17. For group 3, the canals will be dried using suitable size of paper points, followed by obturation using single cone technique using AH plus as a sealer.
18. Final restoration will be placed.
19. Post-operative pain will be accessed using The Visual Analogue Scale (VAS), after 6, 24, 48, 72 hours, and 7 days. Any analgesic pills taken by the patient will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular molars diagnosed with symptomatic irreversible pulpitis.

Exclusion Criteria:

1. Medically compromised patients.
2. Pregnant patients.
3. Teeth with immature apex formation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
The level of post-endodontic pain | 6 hours
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10 cm with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be)
The level of post-endodontic pain | 24 hours
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10 cm with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be)
The level of post-endodontic pain | 48 hours
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10 cm with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be)
The level of post-endodontic pain | 72 hours
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10 cm with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be)
The level of post-endodontic pain | 7 days
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10 cm with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates